CLINICAL TRIAL: NCT03562234
Title: The CLiFF Study: A Prospective Evaluation of Change in Liver Function and Fat in Patients With Colorectal Liver Metastases Undergoing Pre-operative Chemotherapy
Brief Title: The CLiFF Study: Change in Liver Function and Fat in Pre-operative Chemotherapy for Colorectal Liver Metastases
Acronym: CLiFF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: The Christie NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); National Institute for Health Research, United Kingdom (Other Government); National Health Service, United Kingdom (Other Government); Humedics GmbH (Industry)
Responsible Party: Principal Investigator, Kat Parmar, Clinical Research Fellow in Surgery & Cancer Research, University of Manchester
Other Study IDs: MD189
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer; Liver Metastasis Colon Cancer; Chemotherapy Effect; Obesity
Keywords: Colorectal Cancer; Colorectal Liver Metastases; Obesity Related Cancer; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-op Chemotherapy for CLM: MR & LiMAx: Patients undergoing pre-operative chemotherapy for colorectal liver metastases being treated at the Christie NHS (National Health Service) Foundation Trust.
  No intervention - participants will continue with standard care. Observation of changes in liver fat and liver function measured by MR (Magnetic Resonance) scan and LiMAx test (Maximum liver capacity).
  Interventions: Diagnostic Test: MR; Diagnostic Test: LiMAx

INTERVENTIONS:
Diagnostic Test: MR — Liver fat (measured as a percentage - hepatic fat fraction) will be measured by Magnetic Resonance imaging
Diagnostic Test: LiMAx — Liver function will be measured using the relatively new CE licenced non-invasive LiMAx (Liver Maximum Capacity) test device, manufactured by Humedics GmbH

SUMMARY:
The CLiFF Study will assess changes in liver function and liver fat in patients with colorectal liver metastases (CLM) undergoing pre-operative chemotherapy before liver resection. There will be no change to the standard treatment for CLM. The change in liver fat will be assessed using novel magnetic resonance techniques and the change in liver function will be measured using a newly-developed fully-licensed breath test to give the most accurate measure of liver function possible.

Understanding if these changes are related or reversible will help to understand the relationship between obesity and cancer. This is an important issue, as obesity is now the second most common cause of cancer worldwide.

DETAILED DESCRIPTION:
Obesity is the second most common cause of cancer in the United Kingdom (UK) and bowel cancer is the third most common cancer. Obesity can increase both the chance of developing bowel cancer and it's progression. Increased liver fat is likely to be important in this process, but it is not easy to measure liver fat accurately without invasive biopsies.

Chemotherapy is often used to treat colorectal liver metastases before surgery. It is known that chemotherapy can increase liver fat and can reduce liver function, however it is not known if these changes are either reversible or related.

Understanding the relationship of these changes and their potential reversibility could help plan the best treatment for colorectal liver metastases and to understand the wider relationship between obesity and cancer.

A Manchester cancer research team have developed new MR (magnetic resonance) scan techniques which are better able to measure liver fat levels without needing invasive biopsies. The researchers also have a newly-developed fully-licensed machine which can measure liver function more accurately by using a breath test (LiMAx test), donated to the team for this study by the manufacturer, Humedics GmbH.

Patients undergoing pre-operative chemotherapy for CLM at the Christie Hospital will be invited to join this study. Their liver fat content will be measured using the new MR techniques and their liver function measured using the LiMAx test. These will be measured before chemotherapy, during chemotherapy, and after they finish. Their normal treatment will remain unchanged. When they undergo liver surgery, the section of removed liver will be analysed for fatty changes to help confirm that the MR scans are accurate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified adenocarcinoma of the colon or rectum with radiological evidence of potentially resectable liver metastases, with no evidence of unresectable non-hepatic metastatic disease.
2. Pre-operative chemotherapy planned using Oxaliplatin-based chemotherapy regimen (including FOLFOX, XELOX and OXCAP regimens
3. Age greater than or equal to 18 years
4. WHO (World Health Organisation) performance status 0, 1 or 2
5. Adequate haematological and hepatic function defined by: Hb ³ 10g/dl, WBC ³ 3.0 x 109/L, ANC ³ 1.5 x 109/L, platelet count ³ 100,000/ mm3, total bilirubin < 30 mmol/L, serum AST, ALT and alkaline phosphatase 5 x upper limit of normal
6. Renal function with creatinine clearance 60 mls/min (for full dose) or 30 ml/min for 50%-dose oxaliplatin
7. Patients must have given written informed consent
8. Any woman of childbearing potential must have a negative pregnancy test prior to enrolment in to the study and must take adequate precautions to prevent pregnancy during treatment

Exclusion Criteria:

1. Presence of a medical or psychiatric condition that impairs their ability to give informed consent
2. Presence of any other serious uncontrolled medical conditions
3. Evidence of unresectable non-hepatic metastatic disease
4. Pregnant or lactating women. Adequate contraception must be used in fertile patients
5. Contra-indications to MR scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented resectable or potentially resectable colorectal cancer liver metastases planned to undergo pre-operative standard care chemotherapy at the Christie NHS Foundation Trust,
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in liver fat (hepatic fat fraction) | 21 weeks
  Change in liver fat (measured as a percentage using MR imaging - the hepatic fat fraction) comparing the baseline pre-chemotherapy measurement at Week 1 with measurements at cessation of chemotherapy (Week 13) and 8 weeks after cessation of chemotherapy (Week 21). The expectation based on relevant literature is that chemotherapy will lead to potentially reversible higher levels of liver fat. Therefore the liver fat measurement (hepatic fat fraction) should be higher at week 13 than at week 1, and if this change is reversible, the liver fat should decrease during the eight weeks following cessation of chemotherapy, resulting in the measurement at Week 21 being lower than week 13.
Change in liver function | 21 weeks
  Change in liver function measured by LiMAx test (Liver Maximum Capacity), comparing the baseline pre-chemotherapy measurement at week 1 with a measurement mid-chemotherapy (week 7), a measurement at cessation of chemotherapy (Week 13) and a measurement 8 weeks after cessation of chemotherapy (week 21). The expectation from relevant literature is that chemotherapy should cause a reversible deterioration in liver function, therefore the measurement at Week 7 should be lower than week 1, with the measurement at Week 13 then being lower again than week 7. If this deterioration in liver function is reversible, potentially within 8 weeks of stopping chemotherapy as suggested in the literature, then the measurement at Week 21 should be higher than both week 7 and week 13.

SECONDARY OUTCOMES:
Change in liver enzymes | 28 weeks
  Change in liver enzymes as measured by routinely collected blood biochemistry investigations taken at baseline (Week 1), during chemotherapy (weeks 3, 5, 7, 9 and 11) at cessation of chemotherapy (week 13), at pre-operative assessment (Week 21) and at post-operative outpatient review (Week 28). The expectation is that if any chemotherapy-related deterioration in liver function is detected by a change in liver enzymes, it will not be detected as well as by the LiMAx assessment, therefore any change from baseline values should be less substantial.
Change in body mass index (BMI) | 21 weeks
  BMI measurements taken from routine physical examinations at baseline (Week 1), during chemotherapy (Weeks 3, 5, 7, 9 and 11), at cessation of chemotherapy (Week 13) and at pre-operative assessment (Week 21). Any change in BMI will be compared to the change in liver fat as assessed by MR scan, to establish if an increase in liver fat is related to an overall change in BMI rather than a localised effect of chemotherapy.
Change in CT-derived anthropometric measurements 1 - Visceral Adipose Tissue (VAT) | 21 weeks
  Anthropometric measurements as taken from routine Computed Tomography (CT) scans performed in at baseline (Week 1), cessation of chemotherapy (Week 13) and pre-operative assessment (Week 21). No additional CT scans will be performed other than those indicated by routine standard care. Visceral adipose tissue (VAT) measurements will be calculated from these routine CT scans by measuring the intra-abdominal fat in a single tomographic slice at the L4-L5 level, expressed in centimeters squared. Any change in the VAT measurement will be compared to the change in liver fat as determined by MR scan, in order to assess if any change in liver fat is related to overall changes in body composition rather than being a localised effect on the liver. The change in liver fat will either follow a similar pattern to the change in VAT if it is a generalised change in body composition, or it will be unrelated if it increases via a different mechanism.
Change in CT-derived anthropometric measurements 2 - Subcutaneous Adipose Tissue (SAT) | 21 weeks
  Anthropometric measurements as taken from routine Computed Tomography (CT) scans performed in at baseline (Week 1), cessation of chemotherapy (Week 13) and pre-operative assessment (Week 21). No additional CT scans will be performed other than those indicated by routine standard care. Subcutaneous adipose tissue (SAT) measurements will be calculated from these routine CT scans by measuring the subcutaneous fat in a single tomographic slice at the L4-L5 level, expressed in centimeters squared. Any change in the SAT measurement will be compared to the change in liver fat as determined by MR scan, in order to assess if any change in liver fat is related to overall changes in body composition rather than being a localised effect on the liver. The change in liver fat will either follow a similar pattern to the change in SAT if it is a generalised change in body composition, or it will be unrelated if it increases via a different mechanism.
Change in CT-derived anthropometric measurements 3 - Muscle Mass | 21 weeks
  Anthropometric measurements as taken from routine Computed Tomography (CT) scans performed in at baseline (Week 1), cessation of chemotherapy (Week 13) and pre-operative assessment (Week 21). No additional CT scans will be performed other than those indicated by routine standard care. Muscle mass measurements will be calculated from these routine CT scans by measuring the skeletal muscle mass in a single tomographic slice at the L4-L5 level, expressed in centimeters squared. Any change in the muscle mass measurement will be compared to the change in liver fat as determined by MR scan, in order to assess if any change in liver fat is related to overall changes in body composition rather than being a localised effect on the liver. The change in liver fat will either follow a similar pattern to the change in muscle mass if it is a generalised change in body composition, or it will be unrelated if it increases via a different mechanism.
Digital histological quantification of hepatic fat | 28 weeks
  Hepatic fat fraction as measured by routine histology reporting of operative specimen following surgery to resect liver metastases. This measurement will be compared to the hepatic fat fraction at the Week 21 MR scan in order to assess accuracy in non-invasive assessment of liver fat.
NAS-CRN grade of steatosis (Non-Alcoholic Steatohepatitis Activity Score Clinical Research Network) | 28 weeks
  The Non-Alcoholic Steatohepatitis Clinical Research Network (NASH CRN) have published a NASH activity score (NAS-CRN score). The score assesses the severity of Non-Alcoholic Fatty Liver Disease and is performed during routine histology reporting on liver specimens. It uses the sum of three components to give a total of 0-8 points: 1) Steatosis (0: < 5%; 1: 5 - 33%; 2: 34 - 66%; 3: > 66%), 2) lobular inflammation (0: none; 1: < 2 foci/20x field; 2: 2 - 4 foci/20x field; 3: > 4 foci/20x field), and 3) ballooning degeneration (0: none; 1: few; 2: many). This objective score includes an assessment of the percentage liver steatosis in the sample, representative of overall percentage liver fat. This steatosis score will be compared to the pre-operative measurement of liver fat as determined by MR scan, in order to cross-check the accuracy of this non-invasive technique for the assessment of liver fat.
Post-operative 30 day mortality | 28 weeks
  Post-operative 30 day mortality as yes/no, as routinely collected during standard care.
Post-operative 30 day complications using Clavien-Dindo classification | 28 weeks
  Post-operative 30 day complications as routinely measured during standard care using the standardised Clavien-Dindo classification. This is a standardised grading system for post-operative complications graded by severity from 1 to 5. 1 represents the most minor complications and 5 represents the most severe complication (death).
Post-operative 30 day complications using the Comprehensive Complication Index (CCI) | 28 weeks
  Post-operative 30 day complications as routinely measured during standard care using the Comprehensive Complication Index (CCI). The CCI is a novel metric of postoperative morbidity, integrating in a single formula all complications by severity, ranging from the best possible outcome of 0 (uneventful course) to the worst possible outcome of 100 (death). This is available via an online calculation tool at: https://www.assessurgery.com/about_cci-calculator/
Post-operative 30 day complications using the International Study Group for Liver Surgery (ISGLS) complications score | 28 weeks
  Post-operative 30 day complications as routinely measured during standard care using the International Study Group for Liver Surgery (ISGLS) complications score. This score classifies post-hepatectomy liver failure (PHLF) into three grades of severity- A, B and C. Grade A is the least severe complication with no symptoms and requiring no treatment, and Grade C is the most sever complication involving multisystem organ failure requiring invasive treatment on the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Prof A G Renehan, PhD FRCS, Study Director — The Christie NHS Foundation Trust, The University of Manchester
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parmar KL, O'Reilly D, Valle JW, Braun M, Naish JH, Williams SR, Lloyd WK, Malcomson L, Cresswell K, Bamford C, Renehan AG. Prospective study of change in liver function and fat in patients with colorectal liver metastases undergoing preoperative chemotherapy: protocol for the CLiFF Study. BMJ Open. 2020 Sep 23;10(9):e027630. doi: 10.1136/bmjopen-2018-027630. PMID 32967864